CLINICAL TRIAL: NCT03596021
Title: Turkish Version of "Toe Walking Scale"
Brief Title: The Turkish Validity and Reliability of "Toe Walking Scale" in Children With Idiopathic Toe Walking
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: BezmialemMT
Record Dates: First submitted 2018-06-01; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Exercise; Rehabilitation; Reliability; Validity
Keywords: exercise; toe walking; scale; reliability; validity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In clinics, many scales have been developed to examine daily living activities and function in children with idiopatic toe walking. "The Idiopatic Toe Walking (ITW)" was developed in 2010 by Cylie M.Williams, contains 21 items which measure medical, birth & developmental history and assessment. The aim of the investigator's study was to investigate translating the ITW scale and using it in clinics reliably and valiably with a Turkish version of ITW in children with idiopatic toe walking.

DETAILED DESCRIPTION:
Demographic information was recorded which are included gender, age, using orthosis, botox/surgical history, use and duration of walkers/child-runner (WCR). The scale was translated into Turkish with the following translation steps. Thirty four children with idiopatic toe walking were included in the study. Internal structure consistency and test-retest reliability were measured for reliability analyses. For each item on the scale, Cronbach's alpha coefficient and item-total score correlations were calculated. The scale was administered for test-retest reliability at baseline and one week later by one rater. Test-retest reliability was assessed by Pearson's correlation test with observational gait analysis and 'co-validity' was investigated, statistically.

ELIGIBILITY:
Inclusion Criteria:

* older than 3 years
* without neurologic, orthopethic or psychiatric illnesses
* still walking on toe

Exclusion Criteria:

* absence of any known medical conditions
* no voluntary to participate
* older than 18 years or younger than 3 years

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: diagnosed with toe walking by the pediatric neurologist and conducted to us.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
TOE WALKING SCALE | First: May 2018 Last: one weeks later
  Toe Walking Scale, was developed in 2010 by Cylie M.Williams, contains 21 items which measure medical, birth & developmental history and assessment. The scoring of the scale with Yes/No/Not Applicable. All items themed demographics, neurogenic, neuromuscular, traumatic, and combined them.

SECONDARY OUTCOMES:
Observational gait analysis | First: May 2018 Last: one weeks later
  Observational gait analysis applied by the video recording method. The method have seen after the recording from physiotherapist. The observer will be scored the video records.

CONTACTS AND LOCATIONS:
Overall Officials: Akın İşcan, Prof, Study Director — Bezmialem Vakif University
Locations (1):
- Müberra Tanrıverdi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No